CLINICAL TRIAL: NCT07109102
Title: Exploring Long-Term Benefits of Eccentric Cycling Exercise on Physiological Responses, Exercise Capacity, and Quality of Life in Patients With Type 2 Diabetes Mellitus
Brief Title: Long-Term Benefits of Eccentric Cycling Exercise in Patients With Type 2 Diabetes Mellitus
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Rabiatul Adawiah Abdul Rahman, Principal Investigator, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: USM/JEPeM/PP/25030323
Record Dates: First submitted 2025-07-29; First posted 2025-08-07 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-07

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
Keywords: Eccentric cycling; eccentric exercise; exercise capacity; quality of life; physiological responses; Type 2 diabetes mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: This study is an open-label, single-centre, parallel-group, three-arm, randomised controlled study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Moderate intensity eccentric cycling (MI-ECC) (Experimental)
  Interventions: Other: Moderate-intensity eccentric cycling
- High intensity eccentric cycling (HI-ECC) (Experimental)
  Interventions: Other: High-intensity eccentric cycling
- Moderate intensity concentric cycling (MI-CON) (Active Comparator)
  Interventions: Other: Moderate-intensity concentric cycling

INTERVENTIONS:
Other: Moderate-intensity eccentric cycling — * This group will perform eccentric cycling exercise twice per week for ten weeks using the Cyclus2 standard eccentric ergometer.
  * The intensity will start at 60% of the peak power output (PPO) of the incremental concentric cycling test.
  * The intensity will progressively increase by 5% of PPO every 2 weeks (60%-80% PPO).
  Other Names: MI-ECC
  Arms: Moderate intensity eccentric cycling (MI-ECC)
Other: High-intensity eccentric cycling — * This group will perform eccentric cycling exercise twice per week for ten weeks using the Cyclus2 standard eccentric ergometer.
  * The intensity will start at 80% of the peak power output (PPO) of the incremental concentric cycling test.
  * The intensity will progressively increase by 5% of PPO every 2 weeks (80%-100% PPO).
  Other Names: HI-ECC
  Arms: High intensity eccentric cycling (HI-ECC)
Other: Moderate-intensity concentric cycling — * This group will perform concentric cycling exercise twice per week for ten weeks using the Lode Excalibur sport ergometer.
  * The intensity will start at 60% of the peak power output (PPO) of the incremental concentric cycling test.
  * The intensity will progressively increase by 5% of PPO every 2 weeks (60%-80% PPO).
  Other Names: MI-CON
  Arms: Moderate intensity concentric cycling (MI-CON)

SUMMARY:
The goal of this interventional study is to evaluate the long-term benefits of eccentric (ECC) cycling exercise on physiological responses, exercise capacity, and quality of life (QoL) in patients with type 2 diabetes mellitus (T2DM). The main questions it aims to answer are:

* What are the effects of ECC cycling compared to concentric (CON) cycling on physiological responses, exercise capacity, and QoL in patients with T2DM?
* What are the differential effects of moderate- and high-intensity ECC cycling compared to CON cycling on physiological responses, exercise capacity, and QoL in patients with T2DM?

Researchers will compare moderate- and high-intensity ECC cycling to CON cycling (conventional cycling) to see if ECC cycling can be a viable alternative or complement to existing exercise protocols for managing T2DM.

Participants will:

* Undergo pre-, mid-, and post-intervention assessment
* Perform either moderate- or high-intensity ECC cycling or moderate intensity CON cycling according to group randomisation by the researcher.
* Start with two familiarisation sessions prior to the actual cycling training.
* Perform cycling exercise twice per week for 10 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male diagnosed with T2DM
* Age 30 - 60 years old
* Height ≥155cm (To ensure proper ergonomics, comfort and safety during cycling)
* HbA1C level between 6-8%
* No resistance exercise for ≤ 3 months before participating in the current study.
* Physical inactivity (moderate to vigorous exercise ≤60 minutes weekly based on International Physical Activity Questionnaires-Short Form (IPAQ-SF))

Exclusion Criteria:

* Acute illness or any foot ulcer, diabetic ulcer, retinopathy, kidney, musculoskeletal, cardiovascular, or neurological disorder that could impair exercise performance or pose a risk to participants during exercise.
* Insulin injection

Ages: 30 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Glycated haemoglobin (HbA1C) | Baseline and post-intervention at 10 weeks
Lipid profile | Baseline and post-intervention at 10 weeks
Maximal voluntary contraction (MVC) | Baseline, mid-intervention (6 weeks), and post-intervention (10 weeks).
  isometric quadriceps peak torque (QPT) and isokinetic QPT
Exercise capacity | Baseline, mid-intervention (6 weeks), and post-intervention (10 weeks)
  6-minute walk test (6-MWT)
13-item Revised Version of Diabetes Quality of Life (RV-DQOL13) | Baseline, mid-intervention (6 weeks), and post-intervention (10 weeks)
  Scores range from 13 to 65, with higher scores reflecting reduced quality of life
Short Form-12 (SF-12) health survey | Baseline, mid-intervention (6 weeks), and post-intervention (10 weeks)
  Scoring ranges from 0 to 100, with higher scores indicating better physical and mental health.

SECONDARY OUTCOMES:
Electromyography (EMG) for muscle activity assessment | Baseline, mid-intervention (6 weeks), and post-intervention (10 weeks)
  To assess quadriceps muscle activity (rectus femoris, vastus medialis oblique, and vastus lateralis) during maximal voluntary contraction.
Blood pressure | Baseline and up to 10 weeks
  systolic blood pressure (SBP), diastolic blood pressure (DBP),
Heart rate | Baseline and up to 10 weeks
Borg Category-Ratio scale (Borg CR-10) | Every cycling training session from week 1 to week 10
  The scale ranges from 0 (nothing at all) to 10 (extremely strong) to represent the participants' subjective feelings of breathlessness and leg fatigue.
Body weight | Baseline, mid-intervention (6 weeks), and post-intervention (10 weeks)
  Body weight in kilograms (kg)
Height | Baseline, mid-intervention (6 weeks), and post-intervention (10 weeks)
  Height in centimeters (cm)
Body mass index (BMI) | Baseline, mid-intervention (6 weeks), and post-intervention (10 weeks)
  BMI is calculated as weight (kg) divided by height (m²).
Body circumference | Baseline, mid-intervention (6 weeks), and post-intervention (10 weeks)
  Measure the waist circumference (WC), hip circumference (HC), and thigh circumference (TC) in centimetres with a measuring tape.
The short version of the physical activity enjoyment scale (PACES-S) | Mid-intervention (6 weeks), and post-intervention (10 weeks)
  Exercise enjoyment will be assessed using a five-point Likert scale (1 = strongly disagree to 5 = strongly agree), with total scores ranging from 4 to 20; higher scores indicate greater enjoyment.

CONTACTS AND LOCATIONS:
Locations (1):
- Cardio and Muscle Function Laboratory, Pusat Perubatan USM Bertam, Kepala Batas, Pulau Pinang, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ansari M, Hardcastle S, Myers S, Williams AD. The Health and Functional Benefits of Eccentric versus Concentric Exercise Training: A Systematic Review and Meta-Analysis. J Sports Sci Med. 2023 Jun 1;22(2):288-309. doi: 10.52082/jssm.2023.288. eCollection 2023 Jun. PMID 37293426
- [Background] Borot L, Pageaux B, Laroche D, Vergotte G, Lepers R, Perrey S. Eccentric cycling involves greater mental demand and cortical activation of the frontoparietal network. Scand J Med Sci Sports. 2024 Jan;34(1):e14517. doi: 10.1111/sms.14517. Epub 2023 Oct 9. PMID 37814520
- [Background] Penailillo L, Blazevich AJ, Nosaka K. Factors contributing to lower metabolic demand of eccentric compared with concentric cycling. J Appl Physiol (1985). 2017 Oct 1;123(4):884-893. doi: 10.1152/japplphysiol.00536.2016. Epub 2017 Jun 29. PMID 28663378
- [Background] Hoppeler H. Moderate Load Eccentric Exercise; A Distinct Novel Training Modality. Front Physiol. 2016 Nov 16;7:483. doi: 10.3389/fphys.2016.00483. eCollection 2016. PMID 27899894
- [Background] Marcus RL, Lastayo PC, Dibble LE, Hill L, McClain DA. Increased strength and physical performance with eccentric training in women with impaired glucose tolerance: a pilot study. J Womens Health (Larchmt). 2009 Feb;18(2):253-60. doi: 10.1089/jwh.2007.0669. PMID 19183097
- [Background] Clos P, Laroche D, Stapley PJ, Lepers R. Neuromuscular and Perceptual Responses to Sub-Maximal Eccentric Cycling. Front Physiol. 2019 Mar 28;10:354. doi: 10.3389/fphys.2019.00354. eCollection 2019. PMID 30984032
- [Background] Penailillo L, Blazevich A, Numazawa H, Nosaka K. Metabolic and muscle damage profiles of concentric versus repeated eccentric cycling. Med Sci Sports Exerc. 2013 Sep;45(9):1773-81. doi: 10.1249/MSS.0b013e31828f8a73. PMID 23475167
- [Background] LaStayo P, Marcus R, Dibble L, Frajacomo F, Lindstedt S. Eccentric exercise in rehabilitation: safety, feasibility, and application. J Appl Physiol (1985). 2014 Jun 1;116(11):1426-34. doi: 10.1152/japplphysiol.00008.2013. Epub 2013 Jul 3. PMID 23823152
- [Background] LaStayo PC, Ewy GA, Pierotti DD, Johns RK, Lindstedt S. The positive effects of negative work: increased muscle strength and decreased fall risk in a frail elderly population. J Gerontol A Biol Sci Med Sci. 2003 May;58(5):M419-24. doi: 10.1093/gerona/58.5.m419. PMID 12730250
- [Background] Kudiarasu C, Rohadhia W, Katsura Y, Koeda T, Singh F, Nosaka K. Eccentric-only versus concentric-only resistance training effects on biochemical and physiological parameters in patients with type 2 diabetes. BMC Sports Sci Med Rehabil. 2021 Dec 20;13(1):162. doi: 10.1186/s13102-021-00384-z. PMID 34930480
- [Background] Julian V, Thivel D, Miguet M, Pereira B, Costes F, Coudeyre E, Duclos M, Richard R. Eccentric cycling is more efficient in reducing fat mass than concentric cycling in adolescents with obesity. Scand J Med Sci Sports. 2019 Jan;29(1):4-15. doi: 10.1111/sms.13301. Epub 2018 Oct 4. PMID 30222208
- [Background] Szucs G, Pipicz M, Szabo MR, Csont T, Torok L, Csonka C. Effect of Eccentric Exercise on Metabolic Health in Diabetes and Obesity. Sports Med Open. 2023 Sep 29;9(1):91. doi: 10.1186/s40798-023-00596-2. PMID 37775653
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/37293426/